CLINICAL TRIAL: NCT05044117
Title: Single-agent Capecitabine as Metronomic Chemotherapy in Locoregionally Advanced Head and Neck Squamous Cell Carcinoma (CMHN)：A Phase III, Multicentre, Randomised Controlled Trial
Brief Title: Single-agent Capecitabine as Metronomic Chemotherapy in LAHNSCC (CMHN)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Fujian Medical University Union Hospital (Other); Guangzhou Panyu Central Hospital (Other); The Central Hospital of Yongzhou (Unknown); The First People's Hospital of Huaihua (Unknown); Hanzhong Central Hospital (Other); Yichang Central People's Hospital (Other); Affiliated Hospital of Guangdong Medical University (Other); Jiangmen Central Hospital (Other); Xiang Yang No.1 Peoples Hospital (Unknown)
Responsible Party: Principal Investigator, Ying Sun, Vice president, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMHN
Record Dates: First submitted 2021-09-04; First posted 2021-09-14 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: head and neck squamous cell carcinoma; locoregionally advanced disease; metronomic capecitabine
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical observation (No Intervention): The standard treatment followed by clinical observation.
- Metronomic capecitabine (Experimental): The standard treatment followed by a maintenance therapy with capecitabine (650 mg/m2 bid, d1-21, q3w) for 1 year.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Capecitabine — Metronomic capecitabine (650 mg/m2 bid, d1-21, q3w) for 1 year
  Arms: Metronomic capecitabine

SUMMARY:
The purpose of this study is to investigate whether the addition of metronomic capecitabine to the standard treatment can improve prognosis in locoregionally advanced head and neck squamous cell carcinoma.

DETAILED DESCRIPTION:
The standard treatment for resectable locoregionally advanced squamous cell carcinoma of the head and the neck (LAHNSCC) is a regimen consisting of radical surgery plus radiotherapy or concurrent chemoradiotherapy. And induction chemotherapy plus radical radiotherapy or concurrent chemoradiotherapy is also recommended for locoregionally advanced squamous cell carcinoma of larynx and hypopharynx. With the extensive application of comprehensive treatment, the 5-year overall survival of LAHNSCC has not reached 50% yet. So, it is urgent to explore a regimen with high efficiency and low toxicity on the basis of existing standard treatment.

Two retrospective studies found that the metronomic use of orally administered fluorouracil drugs following the reference treatment significantly improved prognosis in LAHNSCC. And capecitabine is one kind of the oral fluorouracil drugs, which has high efficiency and low toxicity. Indeed, metronomic capecitabine maintenance was shown to be effective in patients with breast cancer, colorectal cancer, and nasopharyngeal carcinoma in phase III trials.

The abovementioned studies suggested the promising use of metronomic capecitabine in LAHNSCC. However, there has been no randomized trials in this field. Therefore, we initiated a randomized phase III trial to investigate the efficacy and safety of the addition of metronomic capecitabine to the standard treatment in LAHNSCC.

ELIGIBILITY:
Inclusion Criteria:

1. Performance status of ECOG grade 0 or 1.
2. Tumor staged as III-IV (as defined by the 8th AJCC edition), with newly histologically confirmed squamous cell carcinoma of oral cavity, oropharynx, larynx or hypopharynx.
3. Complete one of the following treatments:

   1. Radical surgery plus radiotherapy or concurrent chemoradiotherapy
   2. Neoadjuvant therapy plus radical radiotherapy or concurrent chemoradiotherapy
   3. Concurrent chemoradiotherapy
4. Postoperative radiotherapy started within 4 to 8 weeks after completion of radical surgery.
5. Within 4 to 8 weeks after completion of the last radiation dose.
6. No clinical evidence of persistent locoregional disease or distant metastases before enrollment.
7. Adequate hematologic (neutrophil count > 1.5×10^9/L, hemoglobin > 90g/L and platelet count > 100×10^9/L), hepatic (alanine aminotransferase, aspartate aminotransferase ≤ 1.5×ULN, bilirubin ≤ 1.5×ULN, alkaline phosphatase ≤ 2.5×ULN) and renal function (creatinine clearance ≥ 50 ml/min).
8. Patients must be appraised of the investigational nature of the study and provide written informed consent.

Exclusion Criteria:

1. p16 positive.
2. Patients who were known to be intolerable or allergic to capecitabine.
3. Illness that would interfere with oral medication, including dysphagia, chronic diarrhea, or ileus.
4. Prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer.
5. Pregnancy or lactation (consider pregnancy test in women of child-bearing age and emphasize effective contraception during the treatment period).
6. Prior surgery, chemotherapy, radiotherapy or other anti-tumor treatments (except diagnostic) to primary tumor or nodes before the standard therapy.
7. Patients who received surgery treatment, biotherapy or immunotherapy during radiotherapy.
8. Patients who are receiving or highly likely to receive other chemotherapy treatment, biotherapy or immunotherapy after radiotherapy.
9. Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose > 1.5×ULN), and emotional disturbance.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2021-10-18 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 2 years
  PFS will be measured from the day of randomization until treatment failure, death from any cause, or the last follow-up visit, whichever occurred first.

SECONDARY OUTCOMES:
Overall survival | 2 years
  OS will be measured from the day of randomization until death due to any cause, or the last follow-up visit.
Distant failure-free survival | 2 years
  DFFS will be measured from the day of randomization until death until distant metastasis, or the last follow-up visit.
Locoregional failure-free survival | 2 years
  LRFFS will be measured from the day of randomization until death until local and/or regional recurrence, or the last follow-up visit.
Adverse events | Up to 2 years
  The incidence of capecitabine-related and other adverse events.
Patient reported quality-of-life score | Up to 2 years
  Patient reported quality of life would be evaluated using the Quality of Life Questionnaire-Core 30 module (QLQ-C30). The score is between 0-100, and the higher score means worse quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Sun, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No